CLINICAL TRIAL: NCT04104490
Title: Angiotensin Converting Enzyme (ACE2), Brain, Gut Dysbiosis in Pulmonary Hypertension
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Mayo Clinic (Other); Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201900896 - N; R01HL102033 (NIH); IRB# 16-001964 (Other: Mayo Clinic); CAAE: 44197015.0.0000.5327 (Other: Federal University of Health Sciences Porto Alegre, Brazil)
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — fecal sample containing microbial DNA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Severe pulmonary arterial hypertension.: This cohort will consist of patients with severe pulmonary arterial hypertension.
  This is defined as mean pulmonary arterial pressure 25 mm Hg or greater and pulmonary artery occlusion pressure 15 mmHg or less measured by right cardiac catheterization and a clinical diagnosis of severe disease.
  Participants will be without signs of left heart disease, lung disease and or hypoxia, chronic thromboembolic pulmonary hypertension or pulmonary hypertension of unclear multifactorial mechanisms.
  This is an observational study with no interventions.
- Mild-moderate pulmonary arterial hypertension: This cohort will consist of patients with mild-moderate pulmonary arterial hypertension.
  This is defined as mean pulmonary arterial pressure 25 mm Hg or greater and pulmonary artery occlusion pressure 15 mmHg or less measured by right cardiac catheterization and a clinical diagnosis of mild-moderate disease.
  Participants will be without signs of left heart disease, lung disease and or hypoxia, chronic thromboembolic pulmonary hypertension or pulmonary hypertension of unclear multifactorial mechanisms.
  This is an observational study with no interventions.
- Reference subjects without pulmonary hypertension: Reference subjects will be healthy people, age- and sex-matched to the other two cohorts, who have no pulmonary artery hypertension.

SUMMARY:
Pulmonary arterial hypertension (PAH) is fatal with right heart failure due to raised pulmonary vascular pressure. Gut dysbiosis was identified in animals with pulmonary hypertension. Deidentified human samples will be tested for gut dysbiosis in PAH, circulating bacterial metabolites and markers of inflammation and gut leakiness. The gut microbiome and circulating metabolites, markers of inflammation and gut leakiness of PAH patients and healthy subjects will be compared in deidentified fecal samples and blood.

DETAILED DESCRIPTION:
Stool samples will be collected from people with no, mild-moderate or severe pulmonary arterial hypertension. Bacterial DNA will be extracted from the feces and sequenced by whole genome sequencing (shotgun sequencing). The DNA sequences will be used to identify the bacteria present in the feces, and to model the functions of the gut microbial community in each of the three groups. This will test for gut dysbiosis in pulmonary arterial hypertensive patients compared to healthy subjects. Gut dysbiosis is a condition where the gut bacterial communities are unbalanced and has been implicated in disease processes.

In subjects recruited in the USA, blood samples will be tested for markers of gut leakiness and inflammation as well as gut bacterial metabolites found in the circulation.

ELIGIBILITY:
Inclusion Criteria:

* severe, mild-moderate or no pulmonary arterial hypertensive subjects

Exclusion Criteria:

* Patients with pulmonary hypertension due to left heart disease, lung diseases and / or hypoxia, chronic thromboembolic pulmonary hypertension, and pulmonary hypertension with unclear multifactorial mechanisms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from pulmonary circulation clinic (Brazil) and the Mayo Clinic (Cardiovascular Division) in Jacksonville, FL
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2015-06-06 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Gut-microbial dysbiosis | 3 weeks
  Identification of fecal microbiota and the function of the gut microbial community

CONTACTS AND LOCATIONS:
Overall Officials: Mohan Raizada, Principal Investigator — University of Florida
Locations (2):
- Mayo Clinic Jacksonville, Jacksonville, Florida, United States
- Universidade Federal de Ciências da Saúde de Porto Alegre, Porto Alegre, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data for primary and secondary outcomes will be made available to other researchers
Supporting Information: Study Protocol
Time Frame: Data will be released a year after completion of the study and or publication of manuscripts containing the data as required by the journal and NIH guidelines.
Access Criteria: The sequence data will be deposited on publicly available sites.